CLINICAL TRIAL: NCT05679817
Title: Effectiveness of a Dose-graded Aerobic Exercise Regimen on Cardiopulmonary Fitness and Physical Performance in Children Survivors of Acute Lymphoblastic Leukemia: A Randomized Clinical Trial
Brief Title: How Effective is the Dose-graded Aerobic Training in Children Survivors of Acute Lymphoblastic Leukemia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0089
Record Dates: First submitted 2022-12-24; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: A prospective, dual-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: A single-blind protocol was adopted. The researcher who collected the data was blind to the allocation of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-GAE group (Experimental): This group received a 12-week aerobic training in addition to the traditional physical rehabilitation.
  Interventions: Other: Dose-graded aerobic exercises
- Control group (Active Comparator): This group received the traditional physical rehabilitation only
  Interventions: Other: Traditional physical rehabilitation

INTERVENTIONS:
Other: Dose-graded aerobic exercises — The D-GAE group received a 12-week aerobic training, three times in addition to the traditional physical rehabilitation. The D-GAE program commenced with a training intensity corresponding to 50% of the maximum age-predicted heart rate for 25 minutes in the first two weeks, which progressed on a two-week basis, and ended up with a training intensity corresponding to 75% of the maximum age-predicted heart rate for 50 minutes in the last two weeks. The D-GAE program included a warm-up for 5 minutes and a cool-down for 5 minutes
  Arms: D-GAE group
Other: Traditional physical rehabilitation — The control group received the traditional physical rehabilitation only, 45 minutes per session, three times a week for 12 consecutive weeks. The program consisted of flexibility exercises, strengthening exercises, balance training, and general conditioning exercises.
  Arms: Control group

SUMMARY:
The purpose of this study was to evaluate the impact of a 12-week dose-graded aerobic exercise program (D-GAE) on cardiopulmonary fitness and physical performance in children survivors of acute lymphoblastic leukemia (ALL). A total of 58 ALL survivors were randomly assigned to the D-GAE group (n = 29, who underwent a combination of traditional physical rehabilitation and intensity- and duration-graded aerobic training three times per week for 12 weeks) or the control group (n = 29, who underwent only traditional physical rehabilitation).

Cardiopulmonary fitness and physical performance were evaluated in both groups before and after treatment.

DETAILED DESCRIPTION:
Fifty-eight survivors of ALL were recruited from the hematology-oncology polyclinic at King Khalid Hospital and two referral pediatric hospitals in Riyadh, Saudi Arabia. The study included survivors aged 10-18 years, who completed maintenance therapy, had no abnormalities of the lower limbs or spine and did not participate in a regular exercise program (in the past six months). survivors who had secondary malignancies, significant musculoskeletal/neurological issues affecting the capacity to participate in exercises or neurocognitive impairments were excluded.

Outcome measures

1. Cardiopulmonary fitness: The peak oxygen uptake was assessed through the McMaster cycling protocol.
2. Physical Performance: Three tests were used; the 6-minute walk test, the timed up and down stairs test, and the 4x10 meter Shuttle Run test.

Interventions

The D-GAE group received a 12-week aerobic training, three times in addition to the traditional physical rehabilitation. The D-GAE program commenced with a training intensity corresponding to 50% of the maximum age-predicted heart rate for 25 minutes in the first two weeks, which progressed on a two-week basis, and ended up with a training intensity corresponding to 75% of the maximum age-predicted heart rate for 50 minutes in the last two weeks. The D-GAE program included a warm-up for 5 minutes and a cool-down for 5 minutes. The control group received the traditional physical rehabilitation only, 45 minutes per session, three times a week for 12 consecutive weeks. The program consisted of flexibility exercises, strengthening exercises, balance training, and general conditioning exercises.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of childhood ALL
* Age of 10-18 years
* Completion of maintenance therapy
* Free of lower limb or spinal deformities
* Not participating in regular exercise regimens in the past six months

Exclusion Criteria:

* Secondary malignancies
* Significant musculoskeletal/neurological issues
* Neurocognitive impairments

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2021-10-03 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake | 3 months
  The peak oxygen uptake (mL/kg/min) was assessed through a symptom-free exercise tolerance test (i.e., the McMaster cycling protocol).

SECONDARY OUTCOMES:
Six-minute walk test. | 3 months
  This test identified the maximum distance (m) that each child was able to cover over six minutes on a straight flat 30-m walkway, without running or jogging. Walking is regarded as more efficient in line with a longer distance coverage
Timed up and down stairs test | 3 months
  This test measured the time (seconds) that each child took to climb up and down a 14-step stair flight (each 20 cm in height). Better performance is indicated by a shorter time.
4x10 meter Shuttle Run test | 3 months
  This test measured the time (seconds) that each child took to run forth and back a 10-meter track. Better performance is indicated by a shorter time.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K. Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No